CLINICAL TRIAL: NCT05848336
Title: Effect of Gluten-free, Casein-free Diet in Children With Autism
Brief Title: The Gluten-Casein-free Diet in Children With Autism: A Clinical Results of the Ophthalmic and Behavioral Manifestations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Mesut Karahan, Assoc. Prof., Uskudar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UskudarUGFCFAUTISM
Record Dates: First submitted 2023-04-26; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder; Ophthalmic Abnormalities
Keywords: gluten free casein free diet
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gluten Free Casein Free Diet (Experimental): Foods containing gluten (pasta, bread, etc.), casein (unfermented dairy products), and their disguised sources have been eliminated from the nutrition program. Also, packaged foods (chocolate, crackers, etc.) containing additives such as artificial preservatives, food coloring, and sweeteners that create a tendency to consume in children were avoided from the nutrition program. Goat milk contains type A2 casein, and most of the casein is digested in fermented dairy products. In order to increase calcium intake, the consumption of some foods (dill, kale, spinach, chard, arugula, broccoli, parsley, legumes, nuts, tahini, etc.) has been increased. Elimination was done gradually, considering nervousness, anxiety, etc., due to the effects of opioid mechanisms of action and gastrointestinal system symptoms.
  Interventions: Behavioral: Gluten Free Casein Free Diet

INTERVENTIONS:
Behavioral: Gluten Free Casein Free Diet — Thirty children with autism were evaluated before the diet (Pre-Test) and after 8 weeks of dietary intervention (Post-Test).

SUMMARY:
To evaluate the efficacy of eight weeks of GFCF in children with ASD on autistic symptoms and ophthalmic findings such as corneal reflex, interpupillary distance (IPD) and pupil size.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a common condition. ASD is a heritable illness characterized by early-onset differences in interaction, communication, sensory atypicality, and stereotyped behaviors. Recent studies suggest a link between elimination diets and severity of autistic behaviors. The etiology of ASD has been still uncertain. Therefore, elucidating the underlying pathology may assist in risk assessment and facilitate process management. Non-harmful and existing evidence for the diet's benefits in ASD must be elucidated.

Primary Study Objective:

To assess the effect of a GFCF diet on variables autism index, stereotyped behaviors, communication, social interaction associated with ASD.

The pupillary response can be utilized to anticipate neurological and physiological activities under the surface. Changes in light trigger the pupil response, which adjusts the amount of brightness falling on the retina by instinctively constricting or dilating the pupil. Atypical pupil size has been linked to abnormal autonomic function in people with ASD. Disturbances in autonomic functions may also lead to differences in the corneal reflex. This study aimed to obtain more data on the behavioral symptoms and ophthalmic measurements of gluten-free casein-free (GFCF) on ASD. In addition, normal development children and children with autism may differ in facial morphology. This study also evaluates the effect of GFCF diet on IPD distance.

Secondary Objectives:

To assess the role of GFCF diet in the manifestation of opthalmic measurements such as pupil size, corneal reflex and IPD.

30 children with ASD were enrolled in a 8-weeks prospective GFCF diet treatment study. In the study, a single group was evaluated with measurements before and after dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent / Assent, as applicable must be signed prior to executing any study related procedure
* Children, male or female, 2 to 11 years old (inclusive)
* Confirmed diagnosis of ASD according to the DSM-IV Symptom Checklist
* Ability to maintain a gluten- and casein-free diet during the study

Exclusion Criteria:

* Cardiovascular, psychiatric, autoimmune, cancer, etc. children with secondary different disease
* Children with any drug use
* Children currently receiving treatment with any alternative medical methods (eg.hyperbaric).
* Children with a diagnosis of celiac disease
* Children who have received any dietary treatment before

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Gilliam Autism Rating Scale 2 (GARS-2) | 8 weeks
  Based on DSM-IV autism diagnostic criteria, GARS-2 is a behavior checklist for children and teenagers aged 3 to 22. The three subscales of the scale are communication, social interaction, and stereotypical behavior. Each subscale contains 14 items that are scored on a four-point scale (0: Never observed, 1: Rarely observed, 2: Sometimes observed, 3: Often observed). The total score obtained from the scale is converted into standard scores, and an OBI score is obtained. An OBI score of 85 and above indicates a high probability of having ASD, a score between 70-84 indicates a medium probability, and a score of 69 and below indicates a low probability.
Weight (kg) | 8 weeks
  Body weight was measured in kilograms.
Body mass index | 8 weeks
  Body mass index (BMI)=weight/(height)^2

SECONDARY OUTCOMES:
The pupil measurements | 8 weeks
  The measurements of both groups were taken from a distance of 1 meter with a binocular photo refractometer under the same conditions, without cycloplegia. Plusoptix® A09 an measure a pupil size of 4.0-8.0 mm in 0.1 mm steps. Eccentric photorefraction is used as a measurement basis. The device provides convenience in terms of pediatric evaluation with its remarkable features. The pupil measurements were performed by an ophthalmologist in the outpatient clinical unit. The brightness level in the room was controlled via the lux meter application. Pupil size (mm) was measured at least three times after each participant was left in a room with a light level of 8 cd/m2 for 2 minutes. The average value of 3 consecutive consistent measurements was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Üsküdar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No